CLINICAL TRIAL: NCT04721418
Title: Aberrant Synaptic Plasticity in Cocaine Use Disorder: A 11C-UCB-J PET Study
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000029552; 1R01DA052454-01A1 (NIH)
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Cocaine Use Disorder; Healthy Controls
MeSH Terms: interventions — 1-((3-(methylpyridin-4-yl)methyl)-4-(3,4,5-trifluorophenyl)pyrrolidin-2-one

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cocaine Use Disorder
  Interventions: Radiation: 11C-UCB-J
- Healthy Control
  Interventions: Radiation: 11C-UCB-J

INTERVENTIONS:
Radiation: 11C-UCB-J — 11C-UCB-J PET scan

SUMMARY:
The purpose of this research study is to measure synaptic density in the brain comparing individuals with cocaine use disorder to healthy controls.

DETAILED DESCRIPTION:
Healthy controls (HC) will be studied as outpatients and undergo one MRI and one 11C-UCB-J PET scan, along with neurocognitive tasks. Individuals with Cocaine Use Disorder (CUD) will complete the study as inpatients on our unit and undergo one MRI and two 11C-UCB-J PET scans, along with neurocognitive tasks. Participants will complete sleep studies (to evaluate sleep architecture); the first two nights after admission and the last two nights before discharge. Cocaine users will be asked to complete outpatient follow-ups twice a week for up to nine weeks following their inpatient stay.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-60 years
* Physically healthy by medical history, physical, neurological, ECG and laboratory examinations
* For females, a negative serum pregnancy test
* For CUD: DSM-5 criteria for Cocaine Use Disorder and positive urine toxicology showing recent use
* For HC: Negative urine toxicology

Exclusion Criteria:

* DSM-5 criteria for other substance use disorders (e.g., alcohol, opiates, sedative hypnotics), except for nicotine
* A primary DSM-5 Axis I major psychiatric disorder (e.g., schizophrenia, bipolar disorder, major depression, etc.) as determined by the Structured Clinical Interview for DSM-5 (SCID-5)
* A history of significant and/or uncontrolled medical or neurological illness
* Current use of psychotropic and/or potentially psychoactive prescription medications
* Medical contraindications to MRI procedure

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: One group will have current Cocaine Use Disorder, the other group will be Healthy Controls
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Between-group (CUD vs. HC) comparisons in ACC. | CUD: After 3 weeks of inpatient abstinence. HC: At baseline as outpatient.
  Between-group comparisons of the fP-corrected total volume of distribution (VT/fP) in ACC.
Between-group (CUD vs. HC) comparisons in vmPFC. | CUD: After 3 weeks of inpatient abstinence. HC: At baseline as outpatient.
  Between-group comparisons of the fP-corrected total volume of distribution (VT/fP) in vmPFC.
Between-group (CUD vs. HC) comparisons in mOFC. | CUD: After 3 weeks of inpatient abstinence. HC: At baseline as outpatient.
  Between-group comparisons of the fP-corrected total volume of distribution (VT/fP) in mOFC.

SECONDARY OUTCOMES:
Within subjects (CUD group) comparisons in ACC. | Baseline versus 3 weeks after.
  Within subjects (CUD group) comparisons (i.e., baseline/pre-abstinence vs. after 3 weeks of inpatient abstinence) of the fP-corrected total volume of distribution (VT/fP) in ACC.
Within subjects (CUD group) comparisons in vmPFC. | Baseline versus 3 weeks after.
  Within subjects (CUD group) comparisons (i.e., baseline/pre-abstinence vs. after 3 weeks of inpatient abstinence) of the fP-corrected total volume of distribution (VT/fP) in vmPFC.
Within subjects (CUD group) comparisons in mOFC. | Baseline versus 3 weeks after.
  Within subjects (CUD group) comparisons (i.e., baseline/pre-abstinence vs. after 3 weeks of inpatient abstinence) of the fP-corrected total volume of distribution (VT/fP) in mOFC.
Between-group (CUD vs. HC) of volume of distribution comparisons in ACC. | CUD: After 3 weeks of inpatient abstinence. HC: At baseline as outpatient.
  Between-group comparisons of volume of distribution (VT) in ACC.
Between-group (CUD vs. HC) of volume of distribution comparisons in vmPFC. | CUD: After 3 weeks of inpatient abstinence. HC: At baseline as outpatient.
  Between-group comparisons of volume of distribution (VT) in vmPFC.
Between-group (CUD vs. HC) of volume of distribution comparisons in mOFC. | CUD: After 3 weeks of inpatient abstinence. HC: At baseline as outpatient.
  Between-group comparisons of volume of distribution (VT) in mOFC.
Between-group (CUD vs. HC) comparisons of binding potential in ACC. | CUD: After 3 weeks of inpatient abstinence. HC: At baseline as outpatient.
  Between-group comparisons of binding potential (BPND) in ACC.
Between-group (CUD vs. HC) comparisons of binding potential in vmPFC. | CUD: After 3 weeks of inpatient abstinence. HC: At baseline as outpatient.
  Between-group comparisons of binding potential (BPND) in vmPFC.
Between-group (CUD vs. HC) comparisons of binding potential in mOFC. | CUD: After 3 weeks of inpatient abstinence. HC: At baseline as outpatient.
  Between-group comparisons of binding potential (BPND) in mOFC.
Between-group (CUD vs. HC) comparisons of gray matter volume in ACC. | CUD: After 3 weeks of inpatient abstinence. HC: At baseline as outpatient.
  Between-group comparisons of gray matter volume (GMV) in ACC.
Between-group (CUD vs. HC) comparisons of gray matter volume in vmPFC. | CUD: After 3 weeks of inpatient abstinence. HC: At baseline as outpatient.
  Between-group comparisons of gray matter volume (GMV) in vmPFC.
Between-group (CUD vs. HC) comparisons of gray matter volume in mOFC. | CUD: After 3 weeks of inpatient abstinence. HC: At baseline as outpatient.
  Between-group comparisons of gray matter volume (GMV) in mOFC.

OTHER OUTCOMES:
Sleep studies | Baseline versus 3 weeks after.
  Investigators will explore the association between synaptic density in the mPFC (measured by VT/fP, with 11C-UCB-J PET) and sleep architecture (measured by slow wave [N3] sleep and total sleep time [TST], using a sleep study device, e.g., polysomnography [PSG]), among subjects with CUD, within 1 week of abstinence and 3 weeks later.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Angarita, MD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States